CLINICAL TRIAL: NCT04717167
Title: The Effect of One Dry Needling Session on Pain and Central Pain Processing in Patients With Knee Osteoarthritis: a Randomized Controlled Trial
Brief Title: The Effect of Dry Needling in Patients With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Sophie Vervullens, Doctoral Candidate, Universiteit Antwerpen
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Supportive Care
Other Study IDs: B3000201630444
Record Dates: First submitted 2021-01-13; First posted 2021-01-20 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Osteoarthritis, Knee
Keywords: dry needling; central pain processing; pain; EMG measurements; muscle coactivation; gait pattern
MeSH Terms: conditions — Osteoarthritis, Knee; Pain | interventions — Dry Needling

STUDY DESIGN:
Intervention Model Description: One group will receive dry needling session and one group will receive placebo treatment. A simple randomization on a website (www.randomizer.org) performed by a researcher (IB), independent from the executive researchers.
Who Masked: Participant, Outcomes Assessor
Masking Description: A double-blinded study was achieved by giving no information about the assigned intervention to the executive researchers; and only the same general explanation about the intervention type to the subjects (Appendix A). Moreover, subjects were prohibited to see the needling-intervention. The group allocation was solely known by the treating therapists and the independent researcher (IB).

ARMS (2):
- DN group (Experimental): All identified MTrPs were inserted with a sterile filiform needle (0,30mm x 40mm or 0,30mm x 75mm, depending on the muscle) that moved up- and downwards until a local twitch response was elicited. When the repeated local twitch response fade away or the subject reported too much pain, the needle was removed. After the treatment, a 15 minutes break(51) was set up and the subjects were not permitted to use a hot pack or to stretch the muscle.
  Interventions: Other: Dry Needling
- Sham needling (SN) group (Sham Comparator): The SN technique was similar to DN, except for penetrating the muscle. In this technique, the needle only penetrated the skin and was therefore impossible to provoke a local twitch response.
  Interventions: Other: Sham Needling

INTERVENTIONS:
Other: Dry Needling
  Arms: DN group
Other: Sham Needling
  Arms: Sham needling (SN) group

SUMMARY:
Research suggests that myofascial trigger points (MTrP) play an important role in explaining pain in patients with musculoskeletal knee disorders. Trigger points are usually defined as hypersensitive tender spots within taut bands of skeletal muscles that are painful on muscle stimulation and that usually elicit referred pain. Treatment of these trigger points could possibly alleviate symptoms in patients with knee pain. However, literature on the effect of trigger point therapy, dry needling in particular, in patients with musculoskeletal knee disorders is scarce. The purpose of this study is to examine the effect of trigger point therapy (dry needling (DN)) on pain, presence of altered central pain processing, muscle features and gait pattern in patients with knee osteoarthritis (KOA). 60 patients with symptomatic KOA will participate in this study. They will randomly be allocated in either an experimental group (EG) (dry needling technique) or a placebo group (PG) (sham needling technique). Pain (Visual analogue scale (VAS) & KOA outcome score (KOOS), muscle features during gait and gait pattern (3D gait analysis and surface electroMyoGraphy (EMG)) and presence of altered central pain processing (Central Sensitization Inventory (CSI), Quantitative Sensory testing (QST)) will be measured at baseline and 15 minutes after the intervention. Additionally, pain will be measured 3 days after the intervention. The investigators hypothesize that the effect on the outcome measures will be significantly larger in the EG compared to the PG.

ELIGIBILITY:
Inclusion Criteria:

* A minimum age of fifty years old;
* Diagnosed with KOA based on the American College of Rheumatology (ACR) clinical classification criteria(48), including:

  * A Kellgren-Lawrence grade of minimum two on radiography;
  * At least three months of chronical knee pain.

Exclusion Criteria:

* Patients suffering from autoimmune and/or neurological disorders
* Patients who had a major trauma/fracture of the lower limb in the past six months -
* Patients who experienced other musculoskeletal problems than OA

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Pain sensation | Change from baseline pain sensation at 15minutes postintervention
  Measured with a Visual Analogue Scale, scored from 0 to 100, where higher scores indicate higher pain sensation.
Pain sensation | Change from baseline pain sensation at 15minutes postintervention
  Measured with the Knee Osteoarthritis Outcome Score- subscale pain, scored on a scale from 0 to 36, transferred from 0 to 100. Higher scores indicate a higher pain sensation.
Pain sensation | Change from baseline pain sensation at 3days postintervention
  Measured with a Visual Analogue Scale, scored from 0 to 100, where higher scores indicate higher pain sensation.
Pain sensation | Change from baseline pain sensation at 3days postintervention
  Measured with the Knee Osteoarthritis Outcome Score- subscale pain, scored on a scale from 0 to 36, transferred from 0 to 100. Higher scores indicate a higher pain sensation.
Pain sensation | Change from 15minutes postintervention pain sensation at 3days postintervention
  Measured with a Visual Analogue Scale, scored from 0 to 100, where higher scores indicate higher pain sensation.
Pain sensation | Change from 15minutes postintervention pain sensation at 3days postintervention
  Measured with the Knee Osteoarthritis Outcome Score- subscale pain, scored on a scale from 0 to 36, transferred from 0 to 100. Higher scores indicate a higher pain sensation.
Pain pressure thresholds | Change from baseline central pain processing at 15minutes postintervention
  Measured with an digital algometer (kilogram force/ square cm)
Temporal summation | Change from baseline central pain processing at 15minutes postintervention
  Measured with an digital algometer (kilogram force/ square cm)
Conditioned pain modulation | Change from baseline central pain processing at 15minutes postintervention
  Measured with an digital algometer (test stimulus) and an inflatable cuff (conditioning stimulus). (kilogram force/ square cm)

SECONDARY OUTCOMES:
Muscle coactivation of musculus Vastus medialis and musculus Semitendinosus | Change from baseline muscle coactivation at 15minutes postintervention
  Measured with wireless surface electromyography. Muscle activation patterns will be gathered through surface electrodes. Hereafter, the co-contraction index was calculated. Higher percentages indicate higher coactivation.
Muscle coactivation of musculus Vastus medialis and musculus Biceps femoris | Change from baseline muscle coactivation at 15minutes postintervention
  Measured with wireless surface electromyography. Muscle activation patterns will be gathered through surface electrodes. Hereafter, the co-contraction index was calculated. Higher percentages indicate higher coactivation.
Muscle coactivation of musculus Vastus lateralis and musculus Semitendinosus | Change from baseline muscle coactivation at 15minutes postintervention
  Measured with wireless surface electromyography. Muscle activation patterns will be gathered through surface electrodes. Hereafter, the co-contraction index was calculated. Higher percentages indicate higher coactivation.
Muscle coactivation of musculus Vastus lateralis and musculus Biceps femoris | Change from baseline muscle coactivation at 15minutes postintervention
  Measured with wireless surface electromyography. Muscle activation patterns will be gathered through surface electrodes. Hereafter, the co-contraction index was calculated. Higher percentages indicate higher coactivation.
Muscle coactivation of musculus Tibialis anterior and musculus Gastrocnemius medialis | Change from baseline muscle coactivation at 15minutes postintervention
  Measured with wireless surface electromyography. Muscle activation patterns will be gathered through surface electrodes. Hereafter, the co-contraction index was calculated. Higher percentages indicate higher coactivation.
Muscle coactivation of musculus Tibialis anterior and musculus Gastrocnemius lateralis | Change from baseline muscle coactivation at 15minutes postintervention
  Measured with wireless surface electromyography. Muscle activation patterns will be gathered through surface electrodes. Hereafter, the co-contraction index was calculated. Higher percentages indicate higher coactivation.
Stride time (seconds) | Change from baseline muscle coactivation at 15minutes postintervention
  measured with force plates and markers to measure toe off and heel strike during a 3D motion analysis.
Stride length (meters) | Change from baseline muscle coactivation at 15minutes postintervention
  measured with force plates and markers to measure toe off and heel strike during a 3D motion analysis.
Step time (meters/second) | Change from baseline muscle coactivation at 15minutes postintervention
  measured with force plates and markers to measure toe off and heel strike during a 3D motion analysis.
Stance phase (%) | Change from baseline muscle coactivation at 15minutes postintervention
  measured with force plates and markers to measure toe off and heel strike during a 3D motion analysis.
Step length (meters) | Change from baseline muscle coactivation at 15minutes postintervention
  measured with force plates and markers to measure toe off and heel strike during a 3D motion analysis.
Step width (meters) | Change from baseline muscle coactivation at 15minutes postintervention
  measured with force plates and markers to measure toe off and heel strike during a 3D motion analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Vervullens, Principal Investigator — Universiteit Antwerpen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vervullens S, Meert L, Baert I, Delrue N, Heusdens CHW, Hallemans A, Van Criekinge T, Smeets RJEM, De Meulemeester K. The effect of one dry needling session on pain, central pain processing, muscle co-contraction and gait characteristics in patients with knee osteoarthritis: a randomized controlled trial. Scand J Pain. 2021 Sep 30;22(2):396-409. doi: 10.1515/sjpain-2021-0091. Print 2022 Apr 26. PMID 34821140